CLINICAL TRIAL: NCT03730168
Title: Response of Inflammatory Markers to Circuit Weight Training in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, assistant professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: p.t.rec/012/001570
Record Dates: First submitted 2018-10-15; First posted 2018-11-05 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus.; Inflammatory markers; Circuit weight training
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group and control group (Experimental): Two groups; study group included 30 diabetic male patients who where trained by circuit weight training program in the form of sets of resistance exercises (in the form of dumbbells and sand bags) for the muscles of lower limb and upper limb .The training sessions were performed 3 days per week for a period of 12 weeks. All patient were on their prescribed routine medications .
  The control group were on there prescribed medications only .
  Interventions: Other: circuit weight training program

INTERVENTIONS:
Other: circuit weight training program — 30 male diabetic patients performed circuit weight training for 12 weeks
  Other Names: Resisted exercises using free weights

SUMMARY:
Study group included 30 male diabetic patients , they performed circuit weight training exercises for 12 weeks in addition to their medications. However, the control group included 10 patients received medical treatment.

Interleukin 6 and tumor necrosis factor alpha were measured before and after the study duration for both groups.

DETAILED DESCRIPTION:
The study group included 30 male diabetic patients who participated in circuit weight training (CWT) program as following; 60 minutes training\day for 3 days per week for a period of 12 weeks.

The training session started by a proper warm up for 5-10 min in the form of mild stretching of the muscles of upper limb(pectorals,shoulder girdle muscles) and muscles of lower limb(flexors, extensors, abductors and adductors of the hip and knee) ( to minimize the risk of musculoskeletal injury). Then start the active phase of resisted exercises through using free weights ( dumbbels for upper limb and sand bags for lower limb) The frequency and intensity increased gradually as follows; Intensity of progress of CWT gradually increased intensity by 2.5% of one repetition maximum every two weeks. Moderate resistance used in which of 60-65% of 1RM in the first month then the intensity increased to 70-75% of 1RM in the second month and finally the intensity of exercises increased to 75-80% of 1RM during the third month. The sets of exercises intervened by 1 min rest in between each set of repetitions. At last the session ends by 10 min of cooling down in the form of relaxation exercises.

Statistical procedures:

In this study, the descriptive statistics (the mean, the standard deviation, maximum, minimum, and range) will be calculated for all subjects in the study including IL6 and tumor necrosis factor alpha variables.

* Paired sample t-test will be used to compare the difference between before and after treatment results of IL6 and tumor necrosis factor alpha in each group.
* Paired T test to compare means of variables before and after training.

ELIGIBILITY:
Inclusion Criteria:

* The selected subjects are diagnosed clinically and laboratory with diabetes mellitus type 2 by physicians.
* All patients have moderate hyperglycemia tested by fasting plasma glucose and a two hours plasma glucose ≥ 200 mg/dl (11.1mmol/l) during an oral glucose tolerance test (OGTT).
* The onset of the disease will be more than 10 years.
* All patients follow an oral hypoglycemicdrug.

Exclusion Criteria:

* Hepatic diseases.
* Cancer patients.
* Renal failure patients.
* Orthopedic problems or fractures of extremities.
* Neurological problems.
* Severely hypertensive patients.

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-13 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
concentration of serum intereukin6 | change from baseline and after 12 weeks
  Laboratory investigation to assess inflammatory marker response to circuit weight training program in male diabetic patients. training was three times weekly for 12 weeks.

SECONDARY OUTCOMES:
concentration of serum tumour necrosis factor | change from baseine and after 12 weeks
  Laboratory investigation to assess inflammatory marker response to circuit weight training program in male diabetic patients. training was three times weekly for 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Cairo Governorate, Egypt